CLINICAL TRIAL: NCT02725606
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Human Serum Albumin/Human Granulocyte-Colony Stimulating Factor(I) Fusion Protein for Injection (GW003) in Patients With Breast Cancer
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of GW003 in Patients With Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-GW003-NP-04
Record Dates: First submitted 2016-03-24; First posted 2016-04-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-01

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Neutropenia; Breast Cancer; GW003
MeSH Terms: conditions — Neutropenia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pegylated Recombinant Human G-CSF (Active Comparator): 100ug/kg 6 subjects (2 subjects per GW003 cohort)
  Interventions: Biological: Pegylated Recombinant Human G-CSF
- GW003 300ug/kg (Experimental): 6-8 subjects
  Interventions: Biological: GW003
- GW003 650ug/kg (Experimental): 6-8 subjects
  Interventions: Biological: GW003
- GW003 850ug/kg (Experimental): 6-8 subjects
  Interventions: Biological: GW003

INTERVENTIONS:
Biological: Pegylated Recombinant Human G-CSF — subcutaneous
  Arms: Pegylated Recombinant Human G-CSF
Biological: GW003 — subcutaneous
  Arms: GW003 300ug/kg; GW003 650ug/kg; GW003 850ug/kg

SUMMARY:
The purpose of the present trial is to evaluate the safety, tolerability and pharmacokinetics(PK)/pharmacodynamics(PD) of single subcutaneous injection of GW003 in breast cancer patients. Moreover, the efficacy will be assessed preliminary.

DETAILED DESCRIPTION:
This is an single-center, open-label, randomized, active-controlled phase I study evaluating tolerability and pharmacokinetics/pharmacodynamics of single subcutaneous injections of GW003 in the breast cancer patients.GW003 is recombinant human serum albumin/human granulocyte-colony stimulating factor(I)fusion protein .It is a long-acting G-CSF(Granulocyte-Colony Stimulating Factor). In this study, participants will be administered a single dose of GW003. Every subject will only accept one dose. In addition to tolerability and safety, pharmacokinetics/pharmacodynamics, preliminary efficacy and immunogenicity of GW003 will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 70 years, female
* Patients with histologically-confirmed breast cancer and plan to accept adjuvant chemotherapy(epirubicin plus cyclophosphamide)
* Have an Eastern Cooperative Oncology Group(ECOG) performance status≤2
* Have no clinically significant impairment in cardiac, liver and kidney
* Adequate hematologic, hepatic and renal function which should meet the following requirements:

  1. Absolute neutrophil count(ANC)≥1.5 x 10^9/L
  2. Blood platelet(PLT)≥100 x 10^9/L
  3. Serum creatinine(sCr)≤1.5 times the upper limit of normal(ULN)
  4. Total bilirubin(TBIL)≤1.5×ULN
  5. Aspartate aminotransferase(AST) /serum glutamic-oxaloacetic transaminase(SGOT) and/or alanine aminotransferase(ALT)/serum glutamic pyruvic transaminase(SGPT) ≤ 2.5 x ULN
  6. Hemoglobin(Hb)>9 g/dL
  7. Alkaline phosphatase(ALP)≤1.5×ULN
* Expected to comply with protocol
* With urine human chorionic gonadotropin (hCG) negative
* Signed informed consent

Exclusion Criteria:

* With acute infection
* With history of bone marrow transplant and/or stem cell transplant
* With primary hematological diseases, such as myelodysplastic syndromes, aplastic anemia, sickle cell anemia
* Received surgery within 3 weeks before chemotherapy
* Received G-CSF within 4 weeks before involved in this study
* Females who are pregnant or lactating
* Participated in other clinical trials at the same time or within 4 weeks before screening
* Known allergy to chemotherapy drugs,recombinant human granulocyte-colony stimulating factor rh(rhG-CSF) or any other biological products
* With cacoethic addiction such as drug abuse or alcoholism
* With other cases which is not suitable for this study judged by investigator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) which are related to GW003 as assessed by CTCAE v4.03 | 21days

SECONDARY OUTCOMES:
Maximum observed maximum plasma concentration [Cmax] | 21days
Time to reach the maximum observed plasma concentration [Tmax] | 21days
Area under the plasma concentration-time curve from time zero to infinity[AUC0-inf] | 21days
Area under the plasma concentration-time curve from time zero to time 't' where t is a defined time point after administration [AUC0-t] | 21days
Terminal elimination half-life[T1/2] | 21days
Absolute neutrophil count[ANC] | 21days
  ANC will be detected pre-dose and 12h,24h,48h,72h,96h,120h,144h,168h,192h,216h,240h,264h,360h,408h,480h post-dose.
CD34+ count | 21days
  CD34+ count will be detected pre-dose and 12h,24h,48h,72h,96h,120h,144h,168h,192h,216h,240h,264h,360h,408h,480h post-dose.
Time to absolute neutrophil count(ANC) recovery | 21days
  The time of ANC of patients who experienced neutropenia after chemotherapy recover to normal levels.
Incidence of severe neutropenia | 21days
  The proportion of patients with grade 3 and 4 neutropenia as assessed by CTCAE v4.03.
Duration of severe neutropenia(DSN) | 21days
  Duration of grade 3 and 4 neutropenia as assessed by CTCAE v4.03.
ANC nadir | 21days
  The minimum value of ANC throughout the study period.
Frequency of subjects with anti-GW003 antibody | 21days
  Anti-GW003 antibody will be detected pre-dose and 21d.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Principal Investigator
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided